CLINICAL TRIAL: NCT04681352
Title: Prospective, Evaluator-blind, Multicenter Study to Assess the Safety and Effectiveness of Treatment With the Octave System for Improving Lines and Wrinkles of the décolleté
Brief Title: A Study of Octave System for Improving Lines and Wrinkles of the Décolleté
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Collaborators: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M960101003
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Results first posted 2023-12-21 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: Décolleté Wrinkles

STUDY DESIGN:
Masking Description: While there was only one arm, Outcome Assessors were masked to pre- vs post-treatment images.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Octave System (Experimental): Single treatment of décolleté tissue.
  Interventions: Device: Octave-Ultherapy treatment

INTERVENTIONS:
Device: Octave-Ultherapy treatment — Micro-focused ultrasound delivered below the surface of the skin.

SUMMARY:
To demonstrate the safety and effectiveness of the Octave System for improving lines and wrinkles of the décolleté.

ELIGIBILITY:
Inclusion Criteria:

- Moderate to severe fine lines, wrinkles, laxity, and crepiness of the décolleté that is amenable to improvement with non-invasive intervention and is not severe enough for surgical intervention.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Scarring in area(s) to be treated.
* Active implants (e.g., pacemakers or defibrillators), ports, or metallic implants in area(s) to be treated.
* Breast implants or is planning to receive breast implants during the study.
* Inability to take pre-treatment medications due to a pre-existing condition, medication allergy, or medical issue that, at the discretion of the treating investigator, is contraindicated.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2022-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.
Locations (10):
- United States (10):
  - Merz Investigational Site #0010395, Beverly Hills, California
  - Merz Investigational Site #0010321, San Mateo, California
  - Merz Investigational Site #0010352, Norwalk, Connecticut
  - Merz Investigational Site #0010416, Miami, Florida
  - Merz Investigational Site #0010346, Chicago, Illinois
  - Merz Investigational Site #0010439, New York, New York
  - Merz Investigational Site #0010452, New York, New York
  - Merz Investigational Site #0010396, Wilmington, North Carolina
  - Merz Investigational Site #0010125, Plano, Texas
  - Merz Investigational Site #0010392, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 10 investigational sites in the United States.
Pre-assignment Details: Of the 153 screened subjects, 54 subjects exited as screen failures and 99 subjects were enrolled to receive a single Octave-Ultherapy treatment in this study.
Groups:
- Octave-Ultherapy Treatment: Subjects received a single Ultherapy treatment with the Octave system on Day 1.
Period: Overall Study
Arm/Group | Octave-Ultherapy Treatment
Started | 99
Completed | 75
Not Completed | 24
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 22

BASELINE CHARACTERISTICS:
Population: The safety population (SP) included all subjects who were enrolled and treated with the Octave System.
Arm/Group | Octave-Ultherapy Treatment
Number analyzed (Participants) | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (6.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 92
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 94
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Treated Subjects With Improvement in Lines and Wrinkles of the Décolleté at Day 90
Description: Improvement in lines and wrinkles of the décolleté were determined after comparing Day 90 photographs with baseline photographs. Improvement was concluded if at least two evaluators assessed the Day 90 photographs as "improved" compared to baseline.
Time Frame: Day 90
Population: Intent-to-treat (ITT) population included all subjects who were enrolled.
Measure: Number; unit: percentage of subjects
Arm/Group | Octave-Ultherapy Treatment
Number analyzed (Participants) | 99
percentage of subjects | 62.2

2. Secondary Outcome: Percentage of Treated Subjects With Improvement in Lines and Wrinkles of the Décolleté at Day 180
Description: Improvement in lines and wrinkles of the décolleté were determined after comparing Day 180 photographs with baseline photographs. Improvement was concluded if at least two evaluators assessed the Day 180 photographs as "improved" compared to baseline.
Time Frame: Day 180
Population: ITT. Here "overall number of subjects analyzed" were subjects who were evaluable for this outcome measure.
Measure: Number; unit: percentage of subjects
Arm/Group | Octave-Ultherapy Treatment
Number analyzed (Participants) | 79
percentage of subjects | 68.0

3. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as adverse events (AEs) with onset or worsening on or after date of first administration of Octave-Ultherapy Treatment.
Time Frame: From Day 1 up to end of the study (Up to Day 180)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Octave-Ultherapy Treatment
Number analyzed (Participants) | 99
Participants | 17

ADVERSE EVENTS:
Time Frame: From Day 1 up to end of the study (Up to Day 180)
Description: Safety Population. The investigator reported AEs systematically at each visit.
Arm/Group | Octave-Ultherapy Treatment
All-Cause Mortality (participants affected / at risk) | 0/99
Serious Adverse Events (participants affected / at risk) | 0/99
Other Adverse Events (participants affected / at risk) | 6/99
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Octave-Ultherapy Treatment (N=99)
Covid-19 (Infections and infestations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Study Protocol (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/52/NCT04681352/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT04681352/SAP_001.pdf